CLINICAL TRIAL: NCT06468761
Title: COVID-19 Infection and 2-year Mortality in Nursing Home Residents Who Survived the First Wave of the Pandemic
Brief Title: 2-year Mortality After COVID-19 in Nursing Home Residents
Status: Completed | Type: Observational
Sponsor: Bichat Hospital (Other)
Responsible Party: Principal Investigator, Manuel Sanchez, Md PhD, Bichat Hospital
Other Study IDs: 22021
Record Dates: First submitted 2024-06-18; First posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Covid19
Keywords: COVID-19; Older Adults; Nursing home; Long-tem mortality
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This was a retrospective study conducted in three Nursing Homes (NHs). Residents who had survived the 1st CoPW (March to May 2020) were included. The diagnosis of COVID-19 was based on the results of a positive reverse transcriptase-polymerase chain reaction test. The collected data also included age, sex, length of residence in the NH, disability status, legal guardianship status, nutritional status, need for texture-modified food, hospitalization or Emergency Department visits during lockdown and SARS-COV2 vaccination status during the follow-up. Non-adjusted and adjusted Cox models were used to analyse factors associated with 2-year post-1stCoPW mortality.

ELIGIBILITY:
Inclusion Criteria:

* Living in one of the Nursing Homes during the fiorst COVID-19 pandemic wave
* Having survived the first pandemic wave

Exclusion Criteria:

* Residents who died during the first pandemic wave
* Refusal for articipation to the study

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: 315 residents of 3 nursibg omes, mean age 86 years old. 50% severe disability. 111 contracted COVID-19 and survived the first pandemic wave.
Sampling Method: Non-Probability Sample
Enrollment: 315 (Actual)
Dates: Start 2020-05-11 (Actual); Primary Completion 2022-07-25 (Actual); Study Completion 2022-07-26 (Actual)

PRIMARY OUTCOMES:
All cause mortality | months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Geriatrics, Paris, France